CLINICAL TRIAL: NCT03316742
Title: Pilot Study on Weight Loss in Guinea Bissau
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has not yet been approved by the local IRB in Guinea Bissau.
Sponsor: Tufts University (Other)
Collaborators: USDA Human Nutrition Research Center on Aging (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Roberts, Director and Senior Scientist, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12377
Record Dates: First submitted 2017-10-13; First posted 2017-10-20 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Overweight and Obesity; Weight Loss
Keywords: Obese; Overweight; Weight loss; West Africa
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention 1 (Experimental): Participants randomized to intervention 1 will complete baseline and endline outcomes and participate in version 1 of a weight loss program. Each participant will attend twelve one hour classes discussing weight loss adherence in addition to barriers experienced. Changes in weight will be recorded throughout the study.
  Interventions: Combination Product: Intervention 1
- Intervention 2 (Experimental): Participants randomized to intervention 2 will complete baseline and endline outcomes and participate in version 2 of a weight loss program. Each participant will attend 12 one hour classes discussing weight loss adherence in addition to barriers experienced. Changes in weight will be recorded throughout the study.
  Interventions: Combination Product: Intervention 2

INTERVENTIONS:
Combination Product: Intervention 1 — Intervention 1 includes providing participants with a high fiber food product, protein source, high intensity sweetener and adult multivitamin.
  Arms: Intervention 1
Combination Product: Intervention 2 — Intervention 2 includes providing participants with an alternative dietary fiber source, milk protein, high intensitysweetener and adult multivitamin.
  Arms: Intervention 2

SUMMARY:
The purpose of this study is to test two versions a weight loss program potentially suitable for implementation in Africa. A successful method would have widespread application in low-income countries, with the potential to improve world health.

DETAILED DESCRIPTION:
Specific Aim 1 is to conduct a 3-4 month pilot study randomizing participants to two versions of a weight loss program. The program will be implemented in a convenience sample of overweight and obese adults living in Guinea-Bissau and measure changes in body weight loss (primary outcome), adherence to program recommendations including recommended food patterns, blood pressure, eating behavior, physical activity and mood (secondary outcomes). The data will be used to refine the weight loss program and conduct power calculations for a future trial.

Specific Aim 2 is to analyze associations between weight loss, participant demographics and program metrics, to explore reasons for differences in weight loss between participants. Factors to be tested include participant BMI, gender and age, as well as adherence to meal portion recommendations, use of sugar-sweetened beverages and provided foods, and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are overweight or obese (BMI ≥25 kg/m2).
* Want to lose weight, want to enroll in the study and are willing to sign the informed consent form.
* Anticipate being able to meet the study requirements for food habits and study meetings, and anticipate remaining in Bissau for the study duration.
* Between the ages of 20 to 65 years.
* Non-pregnant women, and those who do not intend on becoming pregnant during the course of the study.
* A doctor or nurse has signed a note approving participant in the weight loss intervention after seeing a copy of the handout with title "Instructions for Bissau Weight Loss Pilot Project", and a copy of his/her approval is given to the research staff.

Exclusion Criteria:

* Report food allergies or intolerance or health conditions that would prevent consumption of provided and recommended foods.
* Participation in another concurrent nutrition research study.
* If premenopausal (<55 years of age), they are pregnant or intend to become pregnant during the course of the study, or are not using a birth control method to prevent pregnancy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Week 1 - week 12
  Primary outcome is weight change between baseline and endline.

SECONDARY OUTCOMES:
Intervention Adherence | week 1 - week 12
  Adherence to the designated intervention will be measured by self-reported dietary intake.
Change in Blood Pressure | baseline, week 12
  A secondary outcome is change in blood pressure between baseline and endline.
Change in self-reported measures of eating behavior. | baseline, week 12
  Self-administered "Three Factor Eating Questionnaire" will be used to capture participants eating behavior between baseline and endline.
Change in self-reported measures of mood. | baseline, week 12
  Self-administered "Profile of Mood States Questionnaire" will be used to capture participants mood between baseline and endline.
Change in self-reported measures of physical activity. | baseline, week 12
  Self-administered "International Physical Activity Questionnaire" will be used to capture participants physical activity between baseline and endline.
Change in self-reported demographics | baseline, week 12
  A self administered demographics survey measures education, occupation, dietary food frequency and food security.
Change in Height | Week 1, week 12
  A secondary outcome is change in height between baseline and endline.

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Roberts, PhD, Principal Investigator — Tufts University
Locations (1):
- International Partnership for Health Development, Bissau, Guinea-Bissau